CLINICAL TRIAL: NCT05054790
Title: A Phase 2 Study of Augmentation Cystoplasty Using an Autologous Neo-Bladder Construct In Subjects With Fibrotic Contracted Bladder
Brief Title: Augmentation Cystoplasty Using an Autologous Neo-Bladder Construct
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076977
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Contracted Bladder
Keywords: Neo-bladder; fibrotic bladder; bladder compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous "Neo-Bladder" Construct (Experimental): All subjects enrolled will have non-neurogenic, fibrotic contracted bladder that is refractory to medical treatment and require augmentation cystoplasty for preventing long-term sequelae (i.e., kidney failure) that result from persistently high intravesical pressure.
  Interventions: Biological: "Neo-Bladder" Construct

INTERVENTIONS:
Biological: "Neo-Bladder" Construct — Subjects will undergo an open full thickness bladder biopsy from which autologous urinary bladder smooth muscle and urothelial cells will be procured and expanded ex vivo. After approximately 5 - 7 weeks, expanded cells will be seeded on a biodegradable scaffold to produce the neo-bladder construct that will be surgically implanted onto an opened native bladder during an augmentation cystoplasty.

SUMMARY:
The purpose of this research study is to find out if autologous "neo-bladder" construct for the treatment of fibrotic and/or contracted bladder can improve bladder compliance and be safe long term. The neo-bladder is like a reservoir or pouch that will be surgically attached to the bladder to assist with urine collection.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-group clinical study. All subjects will have non-neurogenic, fibrotic contracted bladder that is refractory to medical treatment and require augmentation cystoplasty for preventing long-term sequelae (i.e., kidney failure) that result from persistently high intravesical pressure. Subjects will undergo an open full thickness bladder biopsy from which autologous urinary bladder smooth muscle and urothelial cells will be procured and expanded ex vivo. After approximately 5 - 7 weeks, expanded cells will be seeded on a biodegradable scaffold to produce the neo-bladder construct that will be surgically implanted onto an opened native bladder during an augmentation cystoplasty. Subjects will be followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with small contracted and/or fibrotic non-neurogenic bladder.
* Small bladder <150cc capacity
* Willing and able to give signed informed consent in English.
* Ability of subject to be successfully trained in clean intermittent catheterization and bladder cycling
* Failure to respond to maximum approve dose of medical therapy (e.g. anticholinergics) or failure to tolerate /contraindication to such agents
* Medical need for bladder augmentation, as defined by the presence of:

  1. Decreased and inadequate bladder compliance with a bladder pressure ≥40 cmH20. OR
  2. New-onset of upper urinary tract changes (hydronephrosis, vesicoureteral reflux) in the last 12 months

Exclusion:

* Neurogenic bladder
* Recent (< 12 months) urological or intraperitoneal surgery or device implantation; recent (<6 month neurologic surgery-brain or spine)
* Any prior bladder augmentation procedure
* Known or suspected limitation to obtaining omentum for implantation procedure (e.g., extensive intraperitoneal adhesions)
* Any contraindication to general anesthesia
* Any contraindication or known anaphylactic or severe systemic reaction to either human blood products or materials of bovine origin
* Human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV), active hepatitis A (HAV) or other known active infection
* Subjects with active tuberculosis (TB) requiring treatment in the past 3 years. Subjects with a current positive (≥5 mm induration for high-risk subjects; otherwise ≥10 mm of induration) purified protein derivative (PPD) test are excluded unless they have completed a full course of treatment for latent TB and have a negative chest x-ray film at enrollment.
* Subjects known to be colonized with either methicillin-resistant staphylococcus aureus (MRSA) or vancomycin-resistant Enterococcus (VRE), or gentamicin-resistant organisms.
* Receipt of blood or blood products for transfusion during the 3 months prior to biopsy
* Immunocompromised subjects or subjects receiving immunosuppressive agents (inhaled corticosteroids and chronic low-dose corticosteroids [≤0.25 mg/kg prednisone or equivalent per day] are permitted).
* Brief pulsed corticosteroids for intermittent symptoms (e.g., asthma) are permitted.
* Known history of hypersensitivity to aminoglycosides or fluoroquinolones.
* History of true allergy to iodine or iodinated x-ray contrast agents
* Use of any investigational product within 3 months
* Prior participation in the study
* Any history of alcohol and/or any drug abuse
* Current incarceration for any reason
* Unwillingness, inability, or unlikely compliance with study related procedures
* Any circumstance in which the investigator deems participation in the study is not in the subject's best interest
* Subjects with an Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) value >3 times the upper limit of normal
* Subjects with an albumin value <3.0 g/dL
* Subjects with a history of an anaphylactic or a severe systemic reaction to the biodegradable polymers glycolic acid (PGA) and lactic-co-glycolic acid (PLGA)
* Subjects with acute or chronic abdominal skin infections and/or acute or chronic inflammatory bowel disease
* Subjects with uncontrolled diabetes, unstable cardiac and/or pulmonary disorders, or bleeding disorders
* Subjects who have received Botulinum Toxin A injections into the bladder within the previous 12 months.
* Female subjects who are pregnant, planning to get pregnant or lactating/breast-feeding.
* Female subjects of child-bearing potential unwilling to practice an effective method of birth control as determined by the investigator (e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy) for duration of the study.

  * If a patient has had a hysterectomy, a bilateral oophorectomy, documented ovarian failure or is older than age 51.5 years and has not had a menstrual period in more than 12 months, they will be considered to be non-childbearing. This will be ascertained from patient interview/self-report, medical records (if necessary) and the investigator's judgment. "Spontaneous menopause," occurs in the United States at a mean age of 51.5 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Bladder Compliance Average | Month 12
  Average bladder capacity as found on Urodynamics results
Average Number of 24 Hour Voids | Month 6
  Per voiding diary
Average Number of 24 Hour Voids | Month 9
  Per voiding diary
Average Number of 24 Hour Voids | Month 12
  Per voiding diary

SECONDARY OUTCOMES:
Change in Bladder Capacity | From Baseline through Month 12
  Shown through urodynamics study
End filling pressure | Baseline, Month 6, Month 9 and Month 12
  At age-related nomogram-derived bladder capacity
Urogenital Distress Inventory-6 Question (UDI-6) | Month 6, Month 9 and Month 12
  Evaluation of urogenital function from self-reported questionnaire. Score ranges from 0-18 with higher score denoting worsening in urogenital function.
Urogenital Distress Inventory-7 Question (UDI-7) | Month 6, Month 9 and Month 12
  Evaluation of urogenital function from self-reported questionnaire. Score ranges from 0-21 with higher score denoting worsening in urogenital function.
Genitourinary Pain Index (GUPI) | Month 6, Month 9 and Month 12
  Evaluation of pain from self-reported questionnaire. Score ranges from 0-45 with a higher score denoting worse symptoms.
Quality of Life (QOL) Questionnaire | Month 6, Month 9 and Month 12
  Self-reported quality of life evaluation. Score ranges from 0-6 with highest score denoting the worst feelings about quality of life.
American Urological Association Symptom Score (AUASS) | Month 6, Month 9 and Month 12
  Self-reported urological symptom assesment. Score ranges from 1-35 with score of 1-7 denoting mild symptoms, 8-19 denoting moderate symptoms and 20-35 denoting severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Evans, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No